CLINICAL TRIAL: NCT07294339
Title: 针刺治疗激素受体阳性乳腺癌患者潮热的随机对照试验研究，A Randomized Controlled Trial of Acupuncture for the Management of Hot Flashes in Patients With Hormone Receptor-Positive Breast Cancer
Brief Title: A Randomized Controlled Trial of Acupuncture for the Management of Hot Flashes in Patients With Hormone Receptor-Positive Breast Cancer
Acronym: ACU-HRBC-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Shu Wang, director of breast center, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PekingUPH-LM2025
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Acupuncture Treatment; Hormone Receptor-Positive Breast Cancer; Hot Flashes
Keywords: Hormone Receptor-Positive Breast Cancer; Hot Flashes; Acupuncture; Randomized Controlled Trial
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endocrine therapy + True acupuncture (Experimental)
  Interventions: Other: True Acupuncture
- Endocrine therapy + Sham acupuncture (Other)
  Interventions: Other: Sham Acupuncture

INTERVENTIONS:
Other: True Acupuncture — Acupoints: Sanyinjiao (SP6), Taixi (KI3), Taichong (LR3), Zusanli (ST36) Frequency: 3 sessions per week, for 8 consecutive weeks (24 sessions total) Procedure: Needles inserted to a depth of 0.5 cun, electrical stimulation at 2 Hz, even reinforcing-reducing manipulation until "Deqi" sensation achieved; needles retained for 30 minutes.
  Arms: Endocrine therapy + True acupuncture
Other: Sham Acupuncture — Points: Non-meridian, non-acupoint sites located 0.5-1 cm lateral to true points Frequency: 3 sessions per week, for 8 consecutive weeks Procedure: Needles inserted superficially (0.2 cun) without manipulation or "Deqi" sensation; 2 Hz electrical stimulation applied for 30 minutes.
  Arms: Endocrine therapy + Sham acupuncture

SUMMARY:
Hot flashes are among the most common and distressing adverse effects experienced by patients receiving endocrine therapy for hormone receptor-positive breast cancer. Hormone replacement therapy (HRT) and non-hormonal medications can alleviate symptoms but are limited by side effects and safety concerns, leading to poor adherence. Acupuncture, a traditional Chinese medical therapy involving percutaneous stimulation of specific acupoints, has shown potential to reduce the frequency and severity of hot flashes with minimal adverse events.

This randomized, parallel-controlled clinical trial aims to evaluate the efficacy and safety of acupuncture in managing hot flashes in postoperative breast cancer patients undergoing endocrine therapy. Sixty eligible patients with stage I-III hormone receptor-positive breast cancer will be randomly assigned in a 1:1 ratio to receive either true acupuncture or sham acupuncture, three times per week for eight weeks, followed by a 16-week follow-up period without acupuncture. Functional magnetic resonance imaging (fMRI) will be employed to explore neural mechanisms underlying acupuncture's effects, alongside assessments of hot flash frequency, quality of life (FACT-B+ES), sleep quality (PSQI), and serum biomarkers related to endocrine and neuropeptide regulation. The results are expected to provide evidence for the efficacy and central mechanisms of acupuncture in managing hot flashes in breast cancer patients.

DETAILED DESCRIPTION:
Background Breast cancer is the most prevalent malignancy among women. Advances in multimodal therapy-including surgery, chemotherapy, radiotherapy, endocrine therapy, and targeted therapy-have significantly improved prognosis and survival. However, endocrine therapy frequently induces vasomotor symptoms such as hot flashes, which severely impair quality of life.

Although hormone replacement therapy (HRT) and non-hormonal pharmacologic agents (e.g., SSRIs, anticonvulsants) can alleviate hot flashes, their safety and tolerability remain major limitations. Therefore, there is an urgent clinical need for safe and effective complementary interventions. Acupuncture has been widely used for symptom management in cancer patients due to its convenience, affordability, and safety. Multiple randomized controlled trials (RCTs) have demonstrated its effectiveness in reducing hot flashes and improving quality of life, with few adverse effects.

Functional magnetic resonance imaging (fMRI) studies further indicate that acupuncture can modulate brain regions related to thermoregulation and endocrine function. However, standardized clinical protocols and neuroimaging-based mechanistic studies for tumor-related hot flashes are still limited.

Study Design

This study adopts a single-center, randomized, parallel-controlled design. A total of 60 eligible patients will be randomly allocated (1:1) into two groups:

Group A (Treatment group): Endocrine therapy + True acupuncture Group B (Control group): Endocrine therapy + Sham acupuncture Randomization will be conducted using SAS 9.4 software (SAS Institute, Cary, NC, USA) with a sealed-envelope method. Allocation will be concealed from researchers responsible for recruitment and treatment. The study duration includes 8 weeks of treatment and 16 weeks of follow-up.

Participants Eligible participants are female patients aged 18-75 years with stage I-III hormone receptor-positive breast cancer, currently undergoing endocrine therapy (e.g., selective estrogen receptor modulators, aromatase inhibitors, CDK4/6 inhibitors, with or without ovarian suppression). Participants must have experienced hot flashes for at least 4 weeks, with ≥14 episodes per week and a mean Hot Flash Composite Score (HFCS) of 3-4.

Other key inclusion criteria include ECOG performance status 0-1 and a life expectancy >6 months.

Exclusion criteria include evidence of metastasis, concurrent chemotherapy or radiotherapy, recent use of medications affecting hot flashes (SSRIs, anticonvulsants), unstable cardiac disease, seizure history, MRI contraindications, recent acupuncture for hot flashes, active infection, pregnancy/lactation, or psychiatric/neurological disorders.

Interventions Group A (True Acupuncture) Acupoints: Sanyinjiao (SP6), Taixi (KI3), Taichong (LR3), Zusanli (ST36) Frequency: 3 sessions per week, for 8 consecutive weeks (24 sessions total) Procedure: Needles inserted to a depth of 0.5 cun, electrical stimulation at 2 Hz, even reinforcing-reducing manipulation until "Deqi" sensation achieved; needles retained for 30 minutes.

Group B (Sham Acupuncture) Points: Non-meridian, non-acupoint sites located 0.5-1 cm lateral to true points Frequency: 3 sessions per week, for 8 consecutive weeks Procedure: Needles inserted superficially (0.2 cun) without manipulation or "Deqi" sensation; 2 Hz electrical stimulation applied for 30 minutes.

Both groups continue standard endocrine therapy throughout the trial.

Outcome Measures Primary Outcome fMRI-based neuroimaging analysis: Brain activation patterns and structural changes will be assessed at baseline, mid-treatment, post-treatment, and follow-up to identify neural correlates of acupuncture response.

Secondary Outcomes Hot Flash Diary (HFRDIS): Frequency, severity, and impact on daily life recorded weekly.

Quality of Life: Functional Assessment of Cancer Therapy-Breast plus Endocrine Symptoms (FACT-B+ES, version 4).

Sleep Quality: Pittsburgh Sleep Quality Index (PSQI). Safety Evaluation: Incidence and severity of adverse events during treatment. Exploratory Outcomes Serum biomarkers: Changes in reproductive and neuroendocrine markers, including FSH, LH, E2, P, T, PRL, 5-HT, and CGRP.

Follow-up All participants will be followed up for 16 weeks after completing acupuncture treatment. At the end of follow-up, participants will undergo fMRI scanning and complete the HFRDIS, FACT-B+ES, and PSQI questionnaires.

Safety Assessment Adverse events will be recorded daily throughout the treatment phase. Criteria for early withdrawal include severe adverse reactions, serious complications, physiologic intolerance, loss to follow-up, or patient withdrawal of consent.

Expected Outcomes This trial will evaluate the clinical efficacy and neural mechanisms of acupuncture in alleviating hot flashes among breast cancer patients undergoing endocrine therapy. The findings are expected to provide high-quality evidence supporting acupuncture as a safe, effective, and mechanism-based complementary therapy, and to guide the development of standardized acupuncture protocols for cancer-related vasomotor symptoms.

ELIGIBILITY:
Inclusion Criteria Female patients aged 18 to 75 years. Histopathologically confirmed breast cancer, currently receiving endocrine therapy (e.g., selective estrogen receptor modulators and/or aromatase inhibitors, CDK4/6 inhibitors), with or without ovarian function suppression, for at least 4 weeks and ongoing at the time of enrollment.

Expected survival time > 6 months. Experiencing persistent hot flashes for at least 4 weeks, with a frequency of ≥14 episodes per week (≥2 per day) during the week prior to enrollment, and a Hot Flash Composite Score (HFCS) of 3-4.

Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1:

0: Fully active, able to carry on all pre-disease performance without restriction;

1. Restricted in physically strenuous activity but ambulatory and able to carry out light work (e.g., housework, office work);
2. Ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours;
3. Capable of only limited self-care; confined to bed or chair more than 50% of waking hours;
4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair;
5. Dead. Willing and able to participate in the study and sign the informed consent form.

Exclusion Criteria Evidence of tumor metastasis, currently undergoing radiotherapy, chemotherapy, or having a planned surgery.

Use of selective serotonin reuptake inhibitors (SSRIs) and/or anticonvulsants or other pharmacologic agents for hot flash management within 4 weeks prior to study entry.

Unstable cardiac disease or myocardial infarction within 6 months prior to study initiation.

Recent initiation or modification of endocrine therapy within 1 week, or planned initiation or modification within 14 weeks.

History or risk of seizure of unclear etiology. Prior acupuncture treatment for hot flashes within 6 months before enrollment. Contraindications to MRI scanning. Pregnant or lactating women. Presence of uncontrolled active infection. Severe psychiatric disorders or family history of psychiatric or neurological diseases.

Withdrawal Criteria Failure to complete acupuncture treatment per protocol, making efficacy evaluation impossible.

Use of medications or treatments during the trial that may affect study outcomes.

Voluntary withdrawal from the study during treatment.

Discontinuation Criteria Serious adverse events, complications, or physiological changes during treatment that make continuation unsafe or impractical.

Loss to follow-up or death after enrollment. Participant's voluntary withdrawal at any stage of treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Hormone Receptor-Positive Breast Cancer patient
Enrollment: 60 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Cranial fMRI Imaging Evaluation and Data Analysis | 4 months
  Functional magnetic resonance imaging (fMRI) of the brain will be performed before, during, and after treatment, as well as at the end of follow-up, to assess changes in brain structural and functional imaging characteristics.

SECONDARY OUTCOMES:
Hot Flash Assessment | 4 months
  Hot flash severity and interference with daily life will be evaluated using the Hot Flash Related Daily Interference Scale (HFRDIS). The frequency of hot flashes during the week prior to each follow-up visit will also be recorded and statistically compared between the two groups.
Quality of Life Assessment | 4 months
  Quality of life will be measured using the Functional Assessment of Cancer Therapy-Breast plus Endocrine Subscale (FACT-B, Version 4). The total scores of all subdomains will be analyzed and compared between groups.
Sleep Quality | 4 months
  Sleep quality will be evaluated using the Pittsburgh Sleep Quality Index (PSQI).

OTHER OUTCOMES:
Exploratory Outcome Measures | 4 months
  Exploratory biomarkers will be assessed in peripheral blood samples, including gonadal hormones - follicle-stimulating hormone (FSH), luteinizing hormone (LH), estradiol (E2), progesterone (P), testosterone (T), and prolactin (PRL) - as well as serotonin (5-HT) and calcitonin gene-related peptide (CGRP).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China